CLINICAL TRIAL: NCT02310061
Title: Lung Water By Ultra-Sound Guided Treatment To Prevent Death and Cardiovascular Complications in High Risk End Stage Renal Disease Patients With Cardiomyopathy (Lust Study)
Brief Title: Lung Water by Ultrasound Guided Treatment in Hemodialysis Patients (The Lust Study).
Acronym: LUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Collaborators: Azienda Ospedaliera Bianchi-Melacrino-Morelli (Other); Universität des Saarlandes (Other); Dr. C.I. Parhon Hospital, Iasi (Unknown); Medical University of Silesia (Other); Hospital Universitari de Bellvitge (Other); Central Hospital, Nancy, France (Other); University Hospital, Strasbourg (Other); Shaare Zedek Medical Center (Other); University Medical Centre Maribor (Other); IASIO Hospital - General Clinic of Kallithea (Unknown); ASL Parma (Unknown); University Hospital, Ioannina (Other); Wroclaw Medical University (Other); C.T.M.R. Saint-Augustin (Unknown); Hospital Ambroise Paré Paris (Other); Centre Hospitalier FH Manhes (Other); Aristotle University Of Thessaloniki (Other); Università degli Studi di Ferrara (Other); Istituto di Fisiologia Clinica CNR (Other)
Responsible Party: Principal Investigator, Carmine Zoccali, MD, FASN, Professor of Nephrology (PG), Istituto di Fisiologia Clinica CNR
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERA-EDTA-01062012
Record Dates: First submitted 2014-10-28; First posted 2014-12-05 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Kidney Failure, Chronic
Keywords: Dialysis; ESRD; lung congestion; heart failure; LW-US
MeSH Terms: conditions — Kidney Failure, Chronic; Heart Failure | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (Placebo Comparator): Standard protocol of fluid management in hemodialysis
  Interventions: Other: Standard protocol of fluid management in hemodialysis
- Active arm (Experimental): Extra-vascular lung water measurements by ultrasound (LW-US)
  Interventions: Procedure: Extra-vascular lung water measurements by ultrasound (LW-US)

INTERVENTIONS:
Procedure: Extra-vascular lung water measurements by ultrasound (LW-US) — It is widely agreed that the high prevalence of patients with LV dysfunction and heart failure and the lack of simple, non-expensive, bedside techniques that may serve to estimate and monitor parameters of central hemodynamics for guiding the prescription of ultrafiltration (UF) and drug treatment is a factor of major clinical relevance. So,in patients allocated to the active arm, nephrologists register pre- and post-dialysis US-B lines whenever considered useful for volume monitoring.
  Other Names: LW-US
  Arms: Active arm
Other: Standard protocol of fluid management in hemodialysis — The intervention consists in applying a standard clinical approach for monitoring/tailoring fluid excess in HD patients.
  Arms: Control arm

SUMMARY:
Volume overload is a leading risk factor for death and cardiovascular events in end stage renal disease patients maintained on chronic dialysis, particularly in those with myocardial ischemia and heart failure which represent a substantial fraction of this population. Early identification of volume overload may prevent cardiovascular sequel in these patients but clinical signs of volume expansion are unsatisfactory to reliably identify patients at risk and to monitor them over time. On the other hand, however reliable, standard techniques for measuring extracellular or circulating (blood) volume do not convey information on fundamental heart function parameters that determine the individual haemodynamic tolerance to volume excess and the response to ultrafiltration, i.e. left ventricular (LV) filling pressure and LV function.

Extra-vascular lung water is critically dependent on these parameters and represents a proxy of both, circulating volume and LV filling pressure and function, and may therefore be a better criterion to identify patients at a higher risk of volume-dependent adverse clinical outcomes and to monitor the effect of therapy aimed at preventing these outcomes. A fast (< 5 min.), easy to learn, simple and non-expensive technique which measures extra-vascular lung water by using standard ultrasound (US) machines has been validated in dialysis patients. Whether systematic measurement of lung water by this technique may translate into better clinical outcomes in End Stage Renal Disease (ESRD) patients has never been tested.

The aim of this randomized clinical trial is that of testing a treatment policy guided by extra-vascular lung water measurements by ultrasound to prevent all-cause death, decompensated heart failure and non-fatal myocardial infarction in high risk dialysis patients with myocardial ischemia (a history of myocardial infarction with or without ST elevation or unstable angina, acute coronary syndrome documented by ECG recordings and cardiac troponins or stable angina pectoris with documented coronary artery disease by prior coronary angiography or ECG) or overt heart failure (NYHA class III-IV).

DETAILED DESCRIPTION:
Randomization procedure: After enrollment, patients will be randomized in 2 groups: treatment and control. The randomization will be performed by centre, with a 1:1 allocation ratio, and it will be communicated by the coordinating centre in Reggio Calabria. An allocation concealment will be observed.

Warning: based on the principle "once randomized, always randomized", if a patient drops out the study he cannot simply be replaced by a new one. New patients must be randomized as well.

Validation of core lab data: The core data to be collected in the LUST project/subprojects should be validated by the following validation centres:

* CORE LUST STUDY DATA Echocardiographic data and US-lung data: Dr. Rosa Sicari and Dr. Luna Gargani, CNR Institute of Clinical Physiology of Pisa, Italy (rosas@ifc.cnr.it).
* ANCILLARY LUST PROJECTS Pulse Wave Velocity data (PWV): Prof. Gerard London, Service d'Hémodialyse, Hôpital F.H. Manhès, Fleury-Mérogis, France (glondon@club-internet.fr).

  24 Ambulatory Blood Pressure Monitoring (ABPM) data: Prof. Francesca Mallamaci, Nephrology, Dialysis and Transplantation Unit and IFC-CNR, Reggio Calabria

Preliminary training on US-B lines measurement is a pre-requisite for Nephrologists and Cardiologists of each participating centre. After training (Skype meeting) an online certification will be released to certify the level of expertise about US-B lines measurements of all LUST study nephrologists and cardiologists.

Each participant centre will upload pertinent studies (echocardiography, 24h ABPM and PWV data) into the LUST website and will timely receive a feedback by the validation centres, whenever needed.

US Lung Scan technique A standard (3.0-MHz) echocardiography probe can be used for this purpose. Examinations should be performed in the supine position. To detect lung water, both sides of the chest should be scanned both in the anterior and lateral part from the second to the fourth (on the right side to the fifth) intercostals spaces, at parasternal, mid clavea, anterio-axillar and mid-axillary lines, as previously described (Am J Cardiol 2004;93:1265-70). An US-B line is a hyperechoic, coherent US bundle at narrow basis going from the pleura to the limit of the screen. These extended lines (also called comets) arise from the pleural line and should be differentiated from short comets' artifacts that may exist in other regions. US-B lines starting from the pleural line can be either localized or scattered to the whole lung and be present either as isolated US-B lines or in groups (with a distance >7 mm between 2 extended comets). The sum of US-B lines produces a score reflecting the extent of LW accumulation. If you do not detect any US-B line, the score is 0.

The investigators warn the physicians participating in the trial about fixed US-B lines, due not to lung water but to fibrosis or inflammatory processes. These comets should be registered but not counted as US-B lines. The cause that underlies these artefacts should be described.

In patients allocated to the active arm of the study, any decision about weight reduction will be taken by Nephrologists only on the basis of pre-dialysis US-scans. However, also post-dialysis US-B lines measurement must be performed and registered. In the active and in the control arm as well, US-scans will be performed by the local cardiologist in coincidence with the echocardiographic study. It is crucial for the purpose of this study that cardiologists keep nephrologists involved in the LUST study blinded with respect to the number of US-B lines of patients of the control group.

Timing

* In patients allocated to the control and the active arms, US-B lines should be performed at baseline and at 6, 12 and 24 months by the local cardiologist, in a non-dialysis day either on a Thursday or on a Friday, depending on the dialysis schedule.
* In patients allocated in the treatment arm, the application of US-B scans should be performed as follows:
* In patients with less than 15 US-B lines, ultrafiltration (UF) will not be modified and the US-B lines monitoring will be performed by the nephrologist at monthly intervals;
* In patients with more than 15 US-B lines (either at baseline or at any of the monthly US-B Lung scans) UF will be performed by scheduling longer and/or additional dialyses (see below). In these patients, monitoring of US pre-dialysis and post-dialysis -B lines will be repeated at least once a week, until the goal is achieved (see next section).
* Furthermore, in patients in the active arm, pre- and post-dialysis US-lung scans can be repeated at discretion of the nephrologist, i.e. whenever he/she believes that it can be useful applying this technique for monitoring the volume status of the patient, for example in a patient with <15 US-B lines who subsequently manifests a rise in body weight or in a patient who develops hypotension or frank hypotensive episodes during dialysis .

In brief, in the treatment group, monitoring is scheduled once a week (before and after dialysis), or even more frequently if the nephrologist believes that a more frequent monitoring may be useful to track the desired UF goal. When the number of US-B lines falls below 15, the measurements will be repeated at monthly intervals.

Weight reduction in patients with more than 15 US-B lines

In patients randomized to the treatment arm and with a number of US-B lines >15, a decrease of dry weight is required to reduce lung water, according to the following scheme derived by a pilot study at the coordinating centre and at the Iasi Nephrology Unit:

* 15-30 US-B lines: decrease dry weight by 300 g over the following week (about 100 g per session)
* 31-40 US-B lines: decrease dry weight by 450 g over the following week (about 150 g per session)
* > 40 US-B lines: decrease dry weight by 600 g over next week (about 200 g per session).

Attempts to lower dry weight according to the previous scheme should continue until the US-B lines goal (<15) is attained. If the patient does not tolerate attempts to decrease dry weight for 2 weeks (i.e. if he/she develops hypotension, cramps and other symptoms) extra haemodialysis sessions should be considered.

If the goal (<15 pre-dialysis US B-lines) is not achieved after 4-6 weeks, or in case the patient does not tolerate UF, drug treatment (carvedilol, ACEi, ARB) intensification or introduction should be considered.

Once the goal is achieved, it is recommended to confirm it by repeating the measurement of US-B lines at least once, for example before the following dialysis.

Warnings:

* In patients in the active arm with initial pre-dialysis US-B lines <15 and in those who achieve this goal thanks to body fluids subtraction who develop cramps and/or symptoms of extracellular volume depletion (low dry weight) the decision of increasing dry weight should be accompanied by close US-B lines monitoring (i.e. every dialysis session until the patient stabilizes).
* In patients with >15 pre-dialysis US-B lines who do not tolerate dry weight decrease due to hypotension and who are on hypotensive/cardioprotective drugs treatment (carvedilol/ACEi) the dose of these drugs should be down-titrated and stopped, if needed. These drugs in these patients should be always given after dialysis (before going to bed, at night) rather than pre-dialysis.

Clinical (pre-dialysis) evaluation of volume status In both groups (treatment and control group), a standard pre-dialysis clinical evaluation of volume status should be done, as it is recommended in good clinical practice. This evaluation should consider blood pressure and change of blood pressure over time, pedal edema, presence/absence of dyspnea, crackles on lung auscultation (see below), body weight gain inter-dialysis and body weight trajectory over time. In the active arm of the study these data should also be formally registered whenever US-B lines measurements are done. In the control group, evaluation of volume status needs to be formally registered only in coincidence of the echocardiographic studies.

The following scale will be used for the evaluation of Crackles :

1. No crackles
2. I am uncertain about the presence of fine crackles
3. Definite fine crackles at lung bases
4. Moderate crackles
5. Bilateral, diffuse crackles

For clinical edema, the following scale will be used:

1. No clinical edema
2. Slight pitting (2 mm depth) with no visible distortion
3. Somewhat deeper pit (4 mm) with no readily detectable distortion
4. Noticeably deep pit (6 mm) with the dependent extremity full and swollen
5. Very deep pit (8 mm) with the dependent extremity grossly distorted

Echocardiographic measurements In both the intervention and control arm, cardiologists involved in the LUST study will perform the echocardiographic measurements at baseline, 6, 12 and 24 months, in a non-dialysis day on a Thursday or on a Friday, depending on the dialysis schedule. These echocardiogram are "research echocardiograms". For this reason, it is fundamental to keep nephrologists blind about the results of these echocardiographic readings.

Nevertheless, nephrologists are allowed to consult a cardiologist (be him the LUST cardiologist or another one) for a "clinical echocardiogram" if and when clinical problems arise which demand the application of echocardiographic studies for diagnostic reasons or for monitoring any underlying cardiac problem.

Detailed information about standardization of echocardiographic study has been prepared by echocardiography validation laboratory (Dr. Rosa Sicari and Dr. Luna Gargani, IFC CNR, Pisa).

Statistical analysis plan A total sample size of 500 patients (250 per group) will be expected to provide approximately 80% power to detect a difference in the primary end point with an assumed type I error rate of .05, 2-sided.Investigators estimate that the 2 year event rate for the composite end point would be 45% in the usual care group and 30% (a 33% risk reduction) in the arm with the lung US-guided intervention. According to protocol, all patients will be followed for 24 months after randomization.

Survival analysis will be performed by the Kaplan-Meier and the Cox regression methods. Missing baseline categorical variables will be replaced with the mean or median value, as appropriate. The effect of the allocation arm on the number of US-B lines will be investigated by Linear Mixed Models (LMM).

The between arms differences in echocardiographic data (secondary end point) will be compared by T-Test, Mann-Whitney test and Linear Model Analysis, as appropriate.

A secondary analysis of the longitudinal evolution of US B lines and the time to the first event and to repeated events will be performed by the Joint Models. All analyses will be based on the principle of intention to treat and will be performed using the SPSS version 24, STATA version 13. The threshold for statistical significance will be 2 sided with a type I error rate of .05.

Long-term effect of the intervention In order to capture any long-term effect of the study intervention, data on vital status and cardiovascular events occurred to all patients alive after the intervention period will be collected for additional 24 months after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Dialysis vintage > 3 months
* A history of myocardial infarction with or without ST elevation or unstable angina, acute coronary syndrome, documented by ECG recordings and cardiac troponins, or stable angina pectoris with documented coronary artery disease by prior coronary angiography or ECG or dyspnoea class III-IV NYHA
* Written consent to take part in the study

Exclusion Criteria:

* Cancer or other advanced non cardiac disease or comorbidity (e.g. end-stage liver failure) imposing a very poor short-term prognosis
* Active infections or relevant inter-current disease
* Inadequate lung scanning and echocardiographic studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of the composite outcome "death, myocardial infarction, heart failure". | All events occurred during 24 months of follow up will be assessed at 2 years after the start of the study. For Time-to-Event analyses, we will consider the time from the first visit to the first occurrence of death, or MI or heart failure.
  Myocardial infarction and heart failure will be defined on the basis of international standard protocols.
  - The following figures we expect to occur in the two study arms:
  Active arm: 30% Control arm: 45%

SECONDARY OUTCOMES:
All-cause hospitalizations | First occurrence of all-cause hospitalization over a follow-up period of 24 months
  Hospitalizations due to any cause
Cardiovascular hospitalizations | First occurrence of cardiovascular hospitalization over a follow-up period of 24 months
  All cardiovascular events requiring hospitalization
Left ventricular mass index (LVMI) | LVMI will be measured by cardiologists at baseline, 6, 12 and 24 months
  LVMI will be measured by Echocardiography.
  We expect the following changes in LVMI between the two study arms:
  Active arm: - 2±11 Control arm: 3±11
Left ventricular ejection fraction (LVEF) | LVEF will be measured by cardiologists at baseline, 6, 12 and 24 months
  Left ventricular ejection fraction will be measured by Echocardiography.
  We expect the following changes in LVEF between the two study arms:
  Active arm: 3±9% Control arm: 0±9%
Diastolic function. | Diastolic function (E/E') will be measured by cardiologists at baseline, 6, 12 and 24 months
  Diastolic function will be assessed by Echocardiography.
  We expect the following changes in E/E' between the two study arms:
  Active arm: -2±6 Control arm: 0±6
Left atrial volume | Left atrial volume (LAV) will be measured by cardiologists at baseline, 6, 12 and 24 months
  Left atrial volume will be measured by Echocardiography.
  We expect the following changes in LAV between the two study arms:
  Active arm: -2±17 Control arm: 4±17

OTHER OUTCOMES:
Patients who die of any cause during the follow-up | All deaths occuring over a follow-up period of 24 months
  Death due to any cause
Patients who develop myocardial infarction during the follow-up | First myocardial infarction occuring over a follow-up period of 24 months
  Myocardial infarction as defined according to international standard.
Patients who develop episodes of decompensated heart failure during the follow-up | First heart failure occuring over a follow-up period of 24 months
  Heart failure as defined according to international standard.
Total number of recurrent episodes of decompensated heart failure | All heart failure episodes occuring over a follow-up period of 24 months
  Heart failure as defined according to international standard.
Total number of recurrent cardiovascular events | All cardiovascular events events occuring over a follow-up period of 24 months
  All cardiovascular events as defined according to international standard.
Analysis of hypotension episodes | All hypotension episodes occuring over a follow-up period of 24 months
  All hypotension episodes
Correlation between repeated measurements of lung comets (by US-B lines) and the combined outcome | All combined outcomes (death, myocardial infarction, decompensated heart failure) occuring over a follow-up period of 24 months
  Analysis by joint models combining linear mixed models and survival analysis
Correlation between repeated measurements of lung comets (by US-B lines) and all cause mortality | All deaths occuring over a follow-up period of 24 months
  Analysis by joint models combining linear mixed models and survival analysis
Correlation between repeated measurements of lung comets (by US-B lines) and myocardial infarction | First myocardial infarction occuring over a follow-up period of 24 months
  Analysis by joint models combining linear mixed models and survival analysis
Correlation between repeated measurements of lung comets (by US-B lines) and decompensated heart failure | First episode of heart failure occuring over a follow-up period of 24 months
  Analysis by joint models combining linear mixed models and survival analysis
Correlation between repeated measurements of lung comets (by US-B lines) and Left Ventricular Mass Index (LVMI) | LVMI will be measured by cardiologists at baseline, 6, 12 and 24 months
  Analysis by linear mixed models
Correlation between repeated measurements of lung comets (by US-B lines) and Left Ventricular Ejection Fraction (LVEF) | LVEF will be measured by cardiologists at baseline, 6, 12 and 24 months
  Analysis by linear mixed models
Correlation between repeated measurements of lung comets (by US-B lines) and Diastolic Function (E/E') | E/E' will be measured by cardiologists at baseline, 6, 12 and 24 months
  Analysis by linear mixed models
Correlation between repeated measurements of lung comets (by US-B lines) and Left Atrial Volume (LAV) | LAV will be measured by cardiologists at baseline, 6, 12 and 24 months
  Analysis by linear mixed models
Effect of allocation arm on Sleep Quality | Sleep quality will be assessed at baseline, 6, 12 and 24 months
  Analysis by linear mixed models of the effect of allocation arm on Sleep Quality assessed by Berlin Questionnaire
Effect of allocation arm on Quality of Life | Quality of life will be assessed at baseline, 6, 12 and 24 months
  Analysis by linear mixed models of the effect of allocation arm on Quality of life assessed by by Short Form health survey (SF36)
Effect of allocation arm on Depression | Depression will be assessed at baseline, 6, 12 and 24 months
  Analysis by linear mixed models of the effect of allocation arm on Depression assessed by Center for Epidemiologic Studies - Depression Scale (CES-D)
Effect of allocation arm on overall performance | Performance will be assessed at baseline, 6, 12 and 24 months
  Analysis by linear mixed models of the effect of allocation arm on overall performance assessed by Karnofsky performance score
Effect of allocation arm on Nutritional Status | Nutritional Status will be assessed by at baseline, 6, 12 and 24 months
  Analysis by linear mixed models of the effect of allocation arm on nutritional status assessed by Subjective Global Assessment (SGA)
Analysis of repeated measurements of lung comets (by US-B lines) over time assessed pre-dialysis | All lung comets measured pre-dialysis over a follow-up period of 24 months
  Pre-dialysis lung comets changes and study outcomes
Analysis of repeated measurements of lung comets (by US-B lines) over time assessed post-dialysis | All lung comets measured post-dialysis over a follow-up period of 24 months
  Post-dialysis lung comets changes and study outcomes
Extended follow-up analysis of the composite outcome "death, myocardial infarction, heart failure". | All events occurred during the 24 months follow-up (trial phase) and during 24 months after the end of the study (observational phase)
  Myocardial infarction and heart failure will be defined on the basis of international standard protocols.
Interaction analysis with extended follow-up data | All events occurred during the 24 months follow-up (trial phase) and during 24 months after the end of the study (observational phase)
  As in the main trial, interaction analyses will be performed with gender, age, diabetes, ischemic heart disease, heart failure, number of US-BL, systolic blood pressure, ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Zoccali, Prof, Principal Investigator — CNR-IBIM and Nephrology Unit, Reggio Calabria
Locations (19):
- France (5):
  - C.T.M.R. Saint Augustin, Bordeaux
  - Hôpital Ambroise Paré (Assistance-Publique Hôpitaux de Paris), Boulogne-Billancourt
  - Hôpital F.H. Manhès, Fleury-Mérogis
  - ALTIR - INSERM CHU de Nancy, Nancy
  - University Hospital Strasbourg, Strasbourg
- Saarland University Medical Centre, Homburg/Saar, Germany
- Greece (3):
  - IASIO Hospital - General Clinic of Kallithea, Athens
  - University Hospital of Ioannina, Ioannina
  - Aristotle University, Thessaloniki
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (4):
  - CNR Institute of Clinical Physiology, Pisa, PI
  - CNR-IFC Clinical Epidemiology of Renal Diseases and Hypertension Unit, Reggio Calabria, RC
  - University of Ferrara, Ferrara
  - ASL Parma, Parma
- Poland (2):
  - Medical University of Silesia in Katowice, Katowice
  - Medical University, Wroclaw
- University Hospital 'Dr C.I. Parhon', Iași, Romania
- University Clinical Centre, Maribor, Slovenia
- Bellvitge's University Hispital, Barcelona, Spain

REFERENCES:
- [Background] Kramer A, Stel V, Zoccali C, Heaf J, Ansell D, Gronhagen-Riska C, Leivestad T, Simpson K, Palsson R, Postorino M, Jager K; ERA-EDTA Registry. An update on renal replacement therapy in Europe: ERA-EDTA Registry data from 1997 to 2006. Nephrol Dial Transplant. 2009 Dec;24(12):3557-66. doi: 10.1093/ndt/gfp519. Epub 2009 Oct 9. PMID 19820003
- [Background] Charra B, Calemard E, Ruffet M, Chazot C, Terrat JC, Vanel T, Laurent G. Survival as an index of adequacy of dialysis. Kidney Int. 1992 May;41(5):1286-91. doi: 10.1038/ki.1992.191. PMID 1614043
- [Background] Sinha AD, Agarwal R. Can chronic volume overload be recognized and prevented in hemodialysis patients? The pitfalls of the clinical examination in assessing volume status. Semin Dial. 2009 Sep-Oct;22(5):480-2. doi: 10.1111/j.1525-139X.2009.00641.x. Epub 2009 Sep 9. No abstract available. PMID 19744155
- [Background] Staub NC. Pulmonary edema. Physiol Rev. 1974 Jul;54(3):678-811. doi: 10.1152/physrev.1974.54.3.678. No abstract available. PMID 4601625
- [Background] Crandall ED, Staub NC, Goldberg HS, Effros RM. Recent developments in pulmonary edema. Ann Intern Med. 1983 Dec;99(6):808-22. doi: 10.7326/0003-4819-99-6-808. PMID 6360001
- [Background] Jambrik Z, Monti S, Coppola V, Agricola E, Mottola G, Miniati M, Picano E. Usefulness of ultrasound lung comets as a nonradiologic sign of extravascular lung water. Am J Cardiol. 2004 May 15;93(10):1265-70. doi: 10.1016/j.amjcard.2004.02.012. PMID 15135701
- [Background] Picano E, Gargani L, Gheorghiade M. Why, when, and how to assess pulmonary congestion in heart failure: pathophysiological, clinical, and methodological implications. Heart Fail Rev. 2010 Jan;15(1):63-72. doi: 10.1007/s10741-009-9148-8. PMID 19504345
- [Background] Picano E, Frassi F, Agricola E, Gligorova S, Gargani L, Mottola G. Ultrasound lung comets: a clinically useful sign of extravascular lung water. J Am Soc Echocardiogr. 2006 Mar;19(3):356-63. doi: 10.1016/j.echo.2005.05.019. PMID 16500505
- [Background] Agricola E, Bove T, Oppizzi M, Marino G, Zangrillo A, Margonato A, Picano E. "Ultrasound comet-tail images": a marker of pulmonary edema: a comparative study with wedge pressure and extravascular lung water. Chest. 2005 May;127(5):1690-5. doi: 10.1378/chest.127.5.1690. PMID 15888847
- [Background] Mallamaci F, Benedetto FA, Tripepi R, Rastelli S, Castellino P, Tripepi G, Picano E, Zoccali C. Detection of pulmonary congestion by chest ultrasound in dialysis patients. JACC Cardiovasc Imaging. 2010 Jun;3(6):586-94. doi: 10.1016/j.jcmg.2010.02.005. PMID 20541714
- [Background] Cice G, Ferrara L, Di Benedetto A, Russo PE, Marinelli G, Pavese F, Iacono A. Dilated cardiomyopathy in dialysis patients--beneficial effects of carvedilol: a double-blind, placebo-controlled trial. J Am Coll Cardiol. 2001 Feb;37(2):407-11. doi: 10.1016/s0735-1097(00)01158-x. PMID 11216954